CLINICAL TRIAL: NCT05460312
Title: Assessment of the Expression and Activity of Protein Kinase A in Prostate Cancer Tissue
Brief Title: Protein Kinase A in Prostate Cancer Tissue.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Ran Katz, Dr. Ran Katz, Head, department of Urology, ziv medical center, Ziv Hospital
Other Study IDs: PKA-prostate
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Prostate Neoplasm; Inflammation; Benign Hyperplasia of Prostate
Keywords: protein kinase A; immunohistochemistry; prostate cancer; prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms; Inflammation; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: prostate biopsy — trans rectal ultrasound guided biopsies of prostate . Biopsy smaples will be referred to staining and western blot analysis.

SUMMARY:
Prostate cancer is the most common malignancy in men. documented risk factors of prostate cancer are age, ethnicity, various genomic mutations and family history of prostate cancer. The cellular mechanisms of malignant transformation are numerous and not completely understood. A possible mechanism is induction of an inflammation resulting in cellular atypia and pre-malignant changes in the affected tissue by inducing a pro-inflammatory response or changes in extra cellular matrix. Protein Kinase A (PKA) is a key stone enzyme in various intra-cellular processes. Various infections' inflammations and malignancies were proved to impact PKA activity. The research hypothesis is that prostate cancer tissue will show a unique profile of PKA activity, regulation and intracellular distribution.

DETAILED DESCRIPTION:
The study will be conducted among men referred to prostate biopsy due to clinical suspicion of malignancy. 100 consecutive patients will undergo prostate biopsies. Biopsies will be taken from both lobes of the prostate (standard protocol) and additional biopsies will be taken according to MRI findings (Fusion biopsies) if relevant. One additional biopsy will be taken from each lobe of the prostate and immediately freezed in -80 Celsius degrees. Routine biopsies will be fixed in formaldehyde and embedded in paraffin and will undergo routine pathological analysis and staining.

Following pathological analysis, paraffin slides will be undergo immunohistochemically staining for PKA, comparing cancerous tissue to normal surrounding tissue. the fresh frozen tissue will undergo western blot analysis for quantitative expression of PKA and its sub units.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Clinical suspicion of prostate cancer
* Referred for biopsy
* Able to sign informed consent.

Exclusion Criteria:

* Previous prostate irradiation
* Chronic prostatitis
* Previous prostate surgery
* Recent urinary tract infection (3 months prior to biopsy).
* Indwelling urinary catheter

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men referred to prostate biopsies.
Study Population: A cohort of 100 consecutive men referred to prostate biopsy due to clinical suspicion of prosatet cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
The distribution of PKA in prostate cancer versus benign tissue | 1 year
  Immunohistochemical staining of paraffin sections of prostatebiopsies for PKA, western blot analysisi of tissue.